CLINICAL TRIAL: NCT03182387
Title: Evaluation du Dosage de l'Amylase Dans le Liquide Broncho Alveolaire Dans le Diagnostic précoce de la Pneumopathie d'Inhalation Infectieuse du Sujet Comateux intubé-ventilé.
Brief Title: Key to Improve DiagNosis in Aspiration Pneumonia
Acronym: KIDNAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2015/38
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Infectious Pneumonia; Coma
Keywords: Bronchoalveolar lavage; amylase assay; aspiration pneumonia
MeSH Terms: conditions — Coma; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the diagnostic performance of amylase assay performed from bronchial alveolar fluid to differentiate aseptic chemical inhalation pneumonitis from an infectious inhalation pneumonitis in comatose patients with intubated ventilation for less than 24 hours.

DETAILED DESCRIPTION:
Validation of the potential diagnostic performance of amylase assay compared to gold standard in diagnosis of infectious inhalation pneumonia of the comatose patient enabling the realization of a multicentric study using this innovative method in a diagnostic strategy with the objective of reducing the consumption of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patient intubated ≤ 24 hours for unconsciousness (stroke, meningitis, drug intoxication, metabolic disorders, epilepticus, cardiac arrest).
* Inhalation table with hypoxemic acute respiratory insufficiency post-consciousness + chest x-ray revealing one or more compatible infiltrates + t °> 38 ° C).
* Age ≥18 years
* Patient affiliated to the social security system.
* No opposition obtained

Exclusion Criteria:

* Immunocompromised patient.
* Cardiorespiratory arrest requiring therapeutic hypothermia.
* Pneumopathy nosocomiale (pneumopathy beginning> 48h after hospital admission).
* Infectious Pneumonia in the previous 30 days.
* Previous hospitalization in the previous 30 days.
* Patient under antibiotic at baseline.
* Bacteremia.
* Mechanical ventilation begun before unconsciousness.
* Report Pa02 / FI02 <80.
* Patient under curatorship and / or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to ICU with mechanical ventilation need.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificityof amylase test. | 5 days after inclusion day
  Amylase culture in bronchoalveolar fluid is compared to gold standard culture

CONTACTS AND LOCATIONS:
Overall Officials: Linda Wittkop, PhD, Study Chair — USMR
Locations (1):
- Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No